CLINICAL TRIAL: NCT01944085
Title: Percutaneous Pin Removal in the Outpatient Clinic - do Children Require Analgesia? A Randomized Controlled Trial
Brief Title: Percutaneous Pin Removal in Children - is Analgesia Necessary?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: percpinremoval
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Elbow Fracture
Keywords: children; supracondylar fracture; pin removal; analgesia; pain score
MeSH Terms: conditions — Elbow Fractures; Agnosia | interventions — Acetaminophen; Ibuprofen; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Acetaminophen (Active Comparator): Acetaminophen was administered 1 hour prior to pin removal (weight dependent dose)
  Interventions: Drug: Acetaminophen
- Ibuprofen (Active Comparator): Ibuprofen was administered 1 hour prior to pin removal (weight dependent dose)
  Interventions: Drug: Ibuprofen
- Vitamin C (Placebo) (Placebo Comparator): Vitamin C was administered 1 hour prior to pin removal (weight dependent dose)
  Interventions: Other: Vitamin C

INTERVENTIONS:
Drug: Acetaminophen — Syrup
  Other Names: Paracetamol; Tylenol
  Arms: Acetaminophen
Drug: Ibuprofen — Syrup
  Other Names: Brufen
  Arms: Ibuprofen
Other: Vitamin C — Syrup
  Other Names: Ascorbic Acid
  Arms: Vitamin C (Placebo)

SUMMARY:
This is a simple randomised clinical trial to study if non-narcotic analgesia reduces the pain score and pulse rate of children who undergo removal of percutaneous pins in the outpatient clinic.

Inclusion criteria:

* 5-12 years of age
* 2 or 3 percutaneous pins in either elbow

Exclusion criteria:

- documented or suspected allergies to acetaminophen, ibuprofen

Patients enrolled in the study are instructed not take additional analgesia prior to the clinic visit (risk of overdosage explained). This is verified by clinic nurses conducting the trial.

At the clinic visit, they are randomized into one of three groups

1. acetaminophen; 2. ibuprofen; or 3. Vitamin C (Placebo).

They are served the 'medication' (weight-appropriate dose) and the pins are removed in the clinic an hour later.

Pain score (Wong-Baker scale) and pulse rate are measured before pin removal, immediately following pin removal, and 10 minutes after pin removal.

The study hypothesis is that non-narcotic analgesia (such as acetaminophen and ibuprofen) do not decrease pain score and pulse rate associated with the pin removal procedure.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* age: 5-12 inclusive
* 2 or 3 percutaneous pins in either elbow

Exclusion Criteria:

* documented or suspected allergies to acetaminophen or ibuprofen

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain Score (0 -10) | 10 minutes after pin removal
  Pain score is measured using the Wong-Baker Scale

SECONDARY OUTCOMES:
Pulse rate | 10 minutes after pin removal
  Pulse rate is measured using a pulse oximeter (Nellcor Puritan Bennett - NPB-40)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Lim, MD, FRCS, Principal Investigator — KK Women's & Children's Hospital, SINGAPORE
Locations (1):
- KK Women's & Children's Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Tay GT, Lokino ES, Ong LL, Abdullah SN, Wong ML, Lim KB. Pain during percutaneous pin removal in children with elbow fractures. J Orthop Surg (Hong Kong). 2012 Dec;20(3):369-70. doi: 10.1177/230949901202000322. PMID 23255649
- [Derived] Lim KB, Tan SS, Abdullah SN, Ong LL, Wong ML, Allen JC. Percutaneous pin removal in the outpatient clinic--do children require analgesia?: a randomized controlled trial. J Bone Joint Surg Am. 2014 Apr 2;96(7):597-602. doi: 10.2106/JBJS.M.00806. PMID 24695927